CLINICAL TRIAL: NCT02824627
Title: Investigating the Impact of Oxytocin on Irritability/Emotional Dysregulation in Children and Adolescents With Disruptive Behavior and Mood Disorders, and the Possible Mediating Role of Amygdala Activity
Brief Title: Oxytocin on Irritability/Emotional Dysregulation of Disruptive Behavior and Mood Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0321-16-FB
Record Dates: First submitted 2016-06-27; First posted 2016-07-06 (Estimated); Results first posted 2022-08-30 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Mood Disorder; Disruptive Behavior Disorders
MeSH Terms: conditions — Mood Disorders; Attention Deficit and Disruptive Behavior Disorders | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin (Experimental): Subjects weighing >40kg will receive a total of 24 IU of oxytocin delivered as 2- 6 IU puffs to each nostril once daily. Subjects weighing < 40kg will receive a total of 12 IU of oxytocin delivered as 1- 6 IU puff to each nostril daily. Subjects will receive 14 to 21 days of daily oxytocin administration.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Subjects weighing>40kg will 2 puffs of placebo to each nostril daily. Subjects weighing <40kg will receive 1 puff per day. Subjects will receive 14-21 days of placebo administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — A growing body of data shows that intra-nasal administration of oxytocin has promise for treating a host of psychiatric disorders. Considerable data indicates that oxytocin reduces amygdala response to negative stimuli in patients with generalized anxiety disorder, borderline personality disorder, and post-traumatic stress disorder. Given that one of the potential underlying neurobiological mechanisms of irritability and emotional dysregulation in pediatric population with disruptive behavior and mood disorder is the hyperactivity of amygdala to negative emotional stimuli, and that oxytocin reduces this, it is critical to determine the extent to which this intervention improves irritability and emotional dysregulation in children and adolescents with disruptive behavior and mood disorders.
  Other Names: Pitocin
  Arms: Oxytocin
Drug: Placebo — Inactive substance administered in volume equivalent to volume administered in active treatment arm.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Irritability and emotional dysregulation are recognized as serious aspects of psychopathology seen in in pediatric psychiatric patients. While various behavioral as well as psychopharmacological interventions have shown some efficacy in improving irritability and emotional dysregulation, there are no data determining the neurobiological mechanism of effect at the neural level. Previous studies have demonstrated that heightened amygdala response to negative emotional stimuli is closely related to irritability and emotional dysregulation in children and adolescents. Also, there are studies showing administration of oxytocin can decrease the heightened amygdala response to negative emotional stimuli across various psychiatric diagnoses. This study is a double-blind randomized trial of oxytocin for irritability and emotional dysregulation in the pediatric population. Neuroimaging modalities of fMRI and MEG are employed to probe the neuro-circuitry changes occurring as a result of the oxytocin intervention, specifically including heightened amygdala response to negative emotional stimuli and dysfunctional fronto-amygdala connectivity. The investigators will also investigate the genetic sequence of the oxytocin receptor in the study participants and its relationship with symptom profile and neural activity changes. Children and adolescents (age 10-18) with a diagnosis of disruptive mood and/or behavior disorders (including Attention Deficit/Hyperactivity Disorder [ADHD], Oppositional Defiant Disorder [ODD], Conduct Disorder [CD], and Disruptive Mood Dysregulation Disorder [DMDD]), and clinically significant levels of irritability and emotional dysregulation as measured by the Affective Reactivity Index Scale (score>/= 4).

2 weeks randomized, double-blind treatment with intranasal oxytocin (24 IU daily, or 12 IU daily if the weight is < 40kg) with assessment of diagnosis, symptom profiles (the Affective Reactivity Index [ARI], Inventory of Callous-Unemotional Trait [ICU], Behavior Assessment System for Children, second version [BASC-2], and Clinical Global Impression [CGI]) and pre- and post-oxytocin treatment neuroimaging (fMRI and MEG). The genetic sample will be obtained via buccal mucosa sampling.

Participants may receive outpatient clinically indicated follow-up care in the UNMC department of psychiatry or other local community agency as appropriate.

DETAILED DESCRIPTION:
1. Clinical assessment

   Standard clinical practice at the outpatient clinic of the department of psychiatry, at University of Nebraska Medical Center involves an initial clinical interview by either a child and adolescent psychiatrist faculty member, a child and adolescent psychiatry clinical fellow, or an advanced practice registered nurse. The clinical interview includes past and current history of psychiatric symptoms/signs, past and current medical history, and past/current social/academic history. Also the current medication (if any) and any medical condition that would have interaction with the psychiatric diagnosis will be reviewed. The child/adolescent will receive the diagnosis of psychiatric syndrome at the end of the assessment sessions.
2. Recruitment to the study

   Participants diagnosed with ADHD/CD/ODD/DMDD and presence of clinically significant irritability and emotional dysregulation at the clinical assessment session will be invited to participate in this study afterwards. Participants who respond to advertisement, after a phone screening session will be also invited.
3. Initial research assessment

   Participants who agreed to be enrolled into the protocol will have the initial research assessment session afterwards. This will be held at the outpatient clinic of the department of psychiatry, at University of Nebraska Medical Center. Participants will receive the Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS), to confirm the diagnosis of ADHD/CD/ODD/DMDD, and to rule out any other psychiatric diagnoses listed in the exclusion criteria. Their IQ will be measured by the Wechsler Abbreviated Scale of Intelligence (2-subtest form). Irritability and emotional dysregulation will be measured by the Affective Reactivity Index (ARI). Only the children and adolescents with diagnoses of ADHD/CD/ODD/DMDD and clinically significant level of irritability/emotional dysregulation (score >4 on the ARI) will be enrolled in the study. CBCL, ICU, RPAQ will be used to measure the symptom profiles and functional impairment of patients with ADHD/CD/ODD/DMDD at the initiation and end point of their study participation.
4. fMRI visit 1

   During the MRI visit 1, participants will receive their first fMRI session immediately before initiation of oxytocin or placebo treatment. The fMRI visit 1 can happen on the same day of the initial research assessment after the initial research assessment is completed.

   The Fearful Expression Processing task

   This is a shortened version of the paradigm previously utilized by our group (Marsh & Blair, 2008). During each trial the participant is asked to decide the gender of the face displayed. The face either demonstrates neutral affect or a morphed intensity of fear (50%, 100% or 150%). A trial involves: the presentation of a face (1500 ms) and then a fixation point (1000 ms). There is one run of this task, with 120 face trials (30 neutral, 30 50% fear, 30 100% fear and 30 150% fear) and 60 fixation point trials. In addition, there are 15 seconds of fixation point trials at the beginning and end of the run. Task duration is 8 minutes.

   The Affective Stroop task

   The affective task used here was an adapted version of the paradigm described in previous work. During each trail the participant is asked to decide how many numbers are displayed on the screen, instead of the value of the number. For congruent trials, the numbers were displayed with the same numerosity and number value (e.g., three 3s). For incongruent trials, the numbers were displayed with different numerosities and number values (e.g., four 3s). The individual numerical stimuli consisted of three, four, five, or six 3s, 4s, 5s, or 6s randomly presented within a 9-point grid. There are an equal number of congruent trials and incongruent trials (48 each for a run). These number pictures were preceded and followed by emotional stimuli pictures consisting of 48 positive, 48 negative, and 48 neutral pictures selected from the International Affective Picture System. A trial involves: the presentation of an emotional stimuli (400ms), a numerical display (400ms), the same emotional stimuli (400ms), and a blank (1300ms). Subject completed two runs, generating 288 picture-trial events (32 in each 9 categories) and 96 fixation points to generate a baseline.
5. MEG visit 1

   MEG visit 1 will take place at the Center for MEG (South Doctors Tower, Ste. 222) on the day of their scheduled study. The MEG visit 1 can happen on the same day of the initial research assessment.

   The Emotional Stroop task

   For the emotional Stroop task (EST), three word lists are prepared, a threat list, a negative list, and a neutral list. Each list contains 30 monosyllabic words. The threat words include things encountered in dangerous situation (e.g. gun), the negative words are negative in valence, but not related to threat (e.g., bad). The neutral words are not threatening nor negative (e.g., tune). The three words lists are equated across lexical features including: length, frequency, orthographic, and phonological neighborhood size. Using the ELP database, the words are also equated on average naming latency, naming accuracy, lexical decision time, and lexical decision accuracy (Balota et al., 2007). The task contains 9 experimental blocks, each consisting of 30 color word naming trials from one of our EST lists. The order of the words within each list is randomized across presentation blocks. Within each trial, participants first view a fixation cross for 1 second, which is replaced by a list item that remains on the screen for 2 seconds. An experimenter codes the participant's response as correct (i.e., correct color identification), incorrect (i.e., did not name a color, named the wrong color, or named the word), or as a noise trial (e.g., the participant coughs, etc.). The items are centered horizontally/vertically on a 43.5 by 35cm screen and positioned at eye-level approximately 110cm from the head. Items are presented in red, blue, or green font, and item color is randomly assigned. Reaction times are measured using a dual-plane accelerometer attached to the lower lip and digitized at 1kHz using a Grass amplifier. Voice onset is determined by a sharp increase in the amplitude of the accelerometer signal, which produces response time accuracy near 1ms.
6. Oxytocin/placebo administration

   If the participants are assigned to the oxytocin treatment arm by randomization, they will be initiated on oxytocin administration after the MRI visit 1 and MEG visit 1. Following previous studies using intranasal oxytocin administration, subjects weighing >40kg will receive a total of 24 IU of oxytocin delivered as 2- 6 IU puffs to each nostril once daily. Subjects weighing <40kg will receive a total of 12 IU of oxytocin delivered as 1- 6 IU puff to each nostril daily. Participants will receive 14 to 21 days of daily oxytocin/placebo administration. After 14 days of oxytocin/placebo administration, participants will be scheduled to have MRI visit 2 and MEG visit 2. After those two visits are completed, participants will stop oxytocin/placebo administration. Participants who are assigned to placebo treatment branch will receive identical bottles and instructions for delivery of all the other ingredients of nasal spray except oxytocin. The instruction and demonstration will be given to the parents or legal guardian as the first administration of the nasal spray done at the clinic by either child and adolescent psychiatrist or advanced practice registered nurse. The daily administration will be done by dispatching either oxytocin or placebo nasal spray to the parents of the participants. The oxytocin and placebo nasal spray will be prepared by the University of Nebraska Medical Center research pharmacist who will be un-blinded to each subject's treatment assignment. The randomization will be done by the department of pharmacology by a computer-programmed randomization procedure.

   The participants will have 2 weekly visits to the clinic. They will be assessed for symptom level, nasal spray tolerance, and assessment of adverse effects. Participants will be initiated on psychiatric treatment if it is indicated by change of their psychiatric condition (such as worsening of psychiatric symptoms). In this case, they will not participate in the study any more.

   After 14 days -21 days of trial and the completion of 2nd scans of MRI/MEG and final research assessment, the participants will terminate their participation in this study.
7. MRI visit 2

   MRI visit 2 is identical for all participants to MRI visit 1 and will occur at least 14 days and no more than after 21 days after MRI visit 1. The final research assessment session can occur the same day of MRI visit 2.
8. MEG visit 2

   MEG visit 2 is identical for all participants to MEG visit 1 and will occur at least 14 days and no more than after 21 days after MEG visit 1. The final research assessment session can occur the same day of MRI visit 2.
9. Final research assessment

Final research assessment session will occur at the outpatient clinic of the department of psychiatry at University of Nebraska Medical Center after the MRI visit 2 and the MEG visit 2. During this session, the child and adolescent psychiatrist and the advanced practice registered nurse who are the investigators of this study will administer follow-up assessment of current symptom severity by ARI, CBCL, ICU, RPAQ, as well as compliance with the treatment and side effects.

Participants will be discharged from the study following the final research assessment, or their request to terminate study participation.

If during the course of the study it is discovered that the participant has a disorder or condition that would disqualify him/her (e.g., unexpected side effect of oxytocin that will necessitate cessation of the treatment or medical compromise that will make it impossible to continue oxytocin treatment), but needs further evaluation, the participant will be immediately referred for further clinical assessment and intervention to an appropriate department of University of Nebraska Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* 10-18 years of age
* A current diagnosis of ADHD, ODD, CD, or DMDD as determined by the Kiddie-SADS, lifetime version
* Clinically significant level of irritability as defined by a score of >/=4 on the Affective Reactivity Index (ARI) (Stringaris et al., 2012)
* If currently on medication, medication treatment must be stable for at least 6 weeks with a stimulant medication, alpha 2 agonist, atomoxetine or antidepressant.

Exclusion Criteria:

* Comorbid psychotic, tic, pervasive developmental, or substance abuse disorders
* Major medical illness that prohibits treatment by oxytocin (e.g., severe liver disease, seizure disorder, metabolic disorder)
* Past history of significant worsening of pre-existing psychiatric symptoms after treatment with oxytocin
* Past history of allergic reaction to oxytocin and its nasal spray product
* History of CNS disease (including history of seizure, epilepsy, CNS tumor, CNS hemorrhage, or serious CNS infection including meningitis or encephalitis)
* Current use of antipsychotic medications and anxiolytics (benzodiazepines and barbiturates).
* A positive urine pregnancy test
* A positive urine drug screen or any history of or currently active diagnosis of substance use disorder
* Wechsler Abbreviated Scale of Intelligence (WASI) (D. Wechsler, 1999) scores < 70
* Metal in body (i.e., hearing aid, cardiac pacemaker, bone plates, braces, non-removable piercings/implants, etc), claustrophobia, or any other condition that would preclude fMRI scanning

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soonjo Hwang, MD, Principal Investigator — Assistant Professor, University of Nebraska Medical Center
Locations (1):
- University of Nebraska Medical Center, Department of Psychiatry, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seok JW, Bajaj S, Soltis-Vaughan B, Lerdahl A, Garvey W, Bohn A, Edwards R, Kratochvil CJ, Blair J, Hwang S. Structural atrophy of the right superior frontal gyrus in adolescents with severe irritability. Hum Brain Mapp. 2021 Oct 1;42(14):4611-4622. doi: 10.1002/hbm.25571. Epub 2021 Jul 20. PMID 34288223

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 28 | 30
Completed | 25 | 27
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (2.2) | 13.8 (1.9) | 13.9 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 17 | 24 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 20 | 21 | 41
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Affective Reactivity Index-Youth [Mean (Standard Deviation); unit: units on a scale] — The Affective Reactivity Index -Youth (ARI-Y) is a 7 item inventory specifically designed to measure irritability and emotional dysregulation as a dimensional construct across psychopathologies in children and adolescents (Stingaris et al., 2012). Scores range from 0-12. Total scores are reported. Higher scores are indicative of more (worse) irritability.
  units on a scale | 6.6 (2.2) | 6.5 (2.7) | 6.6 (2.4)
Affective Reactivity Index- Parent [Mean (Standard Deviation); unit: units on a scale] — The Affective Reactivity Index-Parent (ARI-P) is a 7 item inventory (parent-report version) specifically designed to measure irritability and emotional dysregulation as a dimensional construct across psychopathologies in children and adolescents (Stringaris et al., 2012). ARI scores range from 0 to 12. Total scores are reported. Higher scores are indicative of more (worse) irritability. We report the change in ARI score as our outcome measure.
  units on a scale | 7.5 (2.7) | 8.7 (2.0) | 8.1 (2.4)
Clinical Global Impression- Severity [Mean (Standard Deviation); unit: units on a scale] — he Clinical Global Impression: Severity scale is a single-item clinician rated measure of the clinician's impression of the degree of illness of the subject in terms of level of irritability from study start to endpoint. Ratings are 1=normal, not ill, 2= borderline ill, 3= minimally ill, 4= moderately ill, 5= markedly ill, 6= severely ill; 7= very severely ill. A single score of 1 to 7 is given at study endpoint for each subject. A higher score indicates worsening of the subject's irritability based on clinician impression.
  units on a scale | 4.4 (0.6) | 4.6 (0.7) | 4.5 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Affective Reactivity Index - Youth (ARI-Y)
Description: The Affective Reactivity Index-Youth (ARI-Y) is a 7 item inventory (youth self-report) specifically designed to measure irritability and emotional dysregulation as a dimensional construct across psychopathologies in children and adolescents (Stringaris et al., 2012). ARI scores range from 0 to 12. Total scores are reported. Higher scores are indicative of more (worse) irritability. We report the change in ARI-Y score as our outcome measure.
Time Frame: baseline and 21 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 25 | 27
score on a scale | -2.9 (2.3) | -0.8 (2.5)

2. Primary Outcome: Clinical Global Impression: Severity
Description: The Clinical Global Impression: Severity scale is a single-item clinician rated measure of the clinician's impression of the degree of illness of the subject in terms of level of irritability from study start to endpoint. Ratings are 1=normal, not ill, 2= borderline ill, 3= minimally ill, 4= moderately ill, 5= markedly ill, 6= severely ill; 7= very severely ill. A single score of 1 to 7 is given at study endpoint for each subject. A higher score indicates worsening of the subject's irritability based on clinician impression.
Time Frame: 21 days (study endpoint)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 25 | 27
score on a scale | 2.72 (0.79) | 3.33 (1.07)

3. Secondary Outcome: Functional MRI (fMRI) BOLD Response Changes
Description: percent change in BOLD response from baseline to study end point
Time Frame: baseline and 21 days
Population: Number of participants who completed 2 scans (baseline and at the end of the study).
Measure: Mean (Standard Deviation); unit: mean percent change
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 22 | 21
mean percent change | -0.045 (0.007) | 0.045 (0.009)

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 21/25 | 25/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=25) | Placebo (N=27)
Drowsiness (General disorders) | 9 (9) | 6 (6)
Headache (Nervous system disorders) | 3 (3) | 8 (8)
Sleep Disturbance (Psychiatric disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Mood Changes (Psychiatric disorders) | 3 (3) | 8 (8)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (2)
Nose bleeding (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Bad taste (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT02824627/Prot_SAP_005.pdf
  • Informed Consent Form (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT02824627/ICF_006.pdf